CLINICAL TRIAL: NCT01041885
Title: Prospective Feasibility, Non-randomized, Single Arm Multicentre, Multinational Interventional Clinical Investigation Using INSTRUCT Therapy for the Repair of Knee Cartilage Defects
Brief Title: INSTRUCT for Repair of Knee Cartilage Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CellCoTec B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 309-019
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Articular Cartilage Lesion of the Knee
Keywords: knee cartilage defect repair; cartilage lesion; autologous chondrocyte; scaffold; INSTRUCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INSTRUCT (Experimental): INSTRUCT scaffold implantation
  Interventions: Device: INSTRUCT

INTERVENTIONS:
Device: INSTRUCT — INSTRUCT PolyActive scaffold implantation

SUMMARY:
The purpose of this study is to investigate whether the INSTRUCT therapy is safe and effective in the treatment of cartilage defects of the knee.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm pilot study designed to investigate the safety and efficacy of the INSTRUCT therapy in the treatment of knee cartilage defects.

All patients who meet eligibility criteria and who consent to participate will undergo the implantation of a biodegradable scaffold seeded with autologous primary chondrocytes and bone marrow cells via arthrotomy.

Patients will be followed-up for 2 years at regular intervals. Evaluations will include adverse events collection, patient reported outcomes (mostly pain and function), arthroscopic and histologic evaluations and MRIs (including dGEMRIC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic articular cartilage defect in the knee

Exclusion Criteria:

* Surgery on the study knee joint within 6 months
* Patients with significant malalignment (more than 5°)
* Patients with ligamentous instability of the knee
* Majority of the meniscus absent
* Severe osteoarthritis
* Intake of medications or treatments having an effect on bone or cartilage formation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of related adverse events | Over 24 months
Lesion filling | 3 months

SECONDARY OUTCOMES:
Incidence of non-related adverse events | 24 months
KOOS, IKDC and pain VAS scores | At all timepoints over 24 months
Histopathology assessments | 6 or 12 months
MRI evaluation of structural repair | Discharge, 3, 6, 12 and 24 months
dGEMRIC assessment of structural repair | 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joël Guidoux, Study Director — CellCoTec B.V.
Locations (6):
- University Hospital Gent, Ghent, Belgium
- Poland (4):
  - University Hospital nber 2 Dr. Jana Biziela, Bydgoszcz
  - NZOZ "Szpital AVIMED" sp. z o.o., Katowice
  - NZOZ Endomedical, Poznan
  - Centrum Medycyny Sportowej (Sports Medicine Center CMS), Warsaw
- Royal Orthopaedic Hospital, Birmingham, United Kingdom

REFERENCES:
- [Derived] Slynarski K, de Jong WC, Snow M, Hendriks JAA, Wilson CE, Verdonk P. Single-Stage Autologous Chondrocyte-Based Treatment for the Repair of Knee Cartilage Lesions: Two-Year Follow-up of a Prospective Single-Arm Multicenter Study. Am J Sports Med. 2020 May;48(6):1327-1337. doi: 10.1177/0363546520912444. Epub 2020 Apr 8. PMID 32267734